CLINICAL TRIAL: NCT03666208
Title: Sirolimus Coated Angioplasty Balloon in the Salvage of Thrombosed Arteriovenous Graft
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCB
Record Dates: First submitted 2018-09-10; First posted 2018-09-11 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: End Stage Renal Failure on Dialysis; Arteriovenous Graft Occlusion

STUDY DESIGN:
Intervention Model Description: This is a phase 2, pilot clinical trial to investigate the effect of SCB on thrombosed AVG. Specifically, we are focusing on AVG as they have a higher thrombosis rate than AVF and the patency rate even after successful thrombolysis is much lower than AVF. As neointimal hyperplasia is the predominant cause for stenosis at the graft vein junction, treatment with Sirolimus will intuitively delay the recurrence of neo-intimal hyperplasia and result in better patency of the AVG after successful thrombolysis.
  Patients with ESRD presenting with a thrombosed AVG between June 2018 and December 2018 will be screened for suitability. Eligible patients of at least 21 years of age will be offered participation. The potential benefits and risks of SCB will be explained and informed consent obtained from participants. A total of 20 patients will be recruited for the trial and they will be followed up for 6 months after the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thrombosed Arteriovenous Graft (Experimental): Single arm pilot study to investigate effect of sirolimus coated balloon in thrombosed arteriovenous graft
  Interventions: Device: Sirolimus Coated Balloon

INTERVENTIONS:
Device: Sirolimus Coated Balloon — Sirolimus has been used in organ transplantation as well as coronary stent due to its antiproliferative properties. It has been proven to has better outcome in animal studies compared to paclitaxel, which is about 22% in the sirolimus group versus 75% re-stenosis rate in paclitaxel group.
  Sirolimus is coated on the surface of the angioplasty balloon and is transferred to the vessel wall when balloon is inflated and in contact with the vessel wall.
  The following table compare sirolimus to paclitaxel. In which sirolimus works by cytostatic mechanism with a ten thousand fold of safety margin. And sirolimus's anti-restenosis effect is optimal with the benefit of lower level of competition and lesser tissue absorption and elution.
  Other Names: Drug eluting device

SUMMARY:
End stage renal disease is on increasing trend. Haemodialysis is the main dialysis modality among these patients which accounts for the incidence of 81.3% in 2015 based on data from Singapore renal registry. Thus, A functioning dialysis vascular access (either arteriovenous Fistula or graft) is critical to the delivery of life-saving haemodialysis treatment to these patients.

The main focus in our study is thrombosed (blocked) AVG as it has higher thrombosis rate and poorer patency rate. Conventionally, to restore the function of the dialysis access, the thrombus (clot) will be lysed with the use of lytic agent; followed by treatment of the underlying stenosis (narrowing) with plain balloon angioplasty (dilatation). However narrowing often recur and multiple repeated angioplasty procedures are needed keep the AVG flowing to prevent clots formation.

Recently developed balloons called drug eluting balloons, are coated with medications to prevent the narrowing from recurring after angioplasty. With these drug balloons, the AVG can potentially continue to have good flow for a longer period of time, hence, decreasing the chance of clotting. A newer generation of drug-eluting balloon, called sirolimus coated balloon, are coated with a medicine called sirolimus. It has been successfully used in the treatment of narrowing of vessels in the leg and heart and it were superior than conventional paclitaxel coated balloon angioplasty.

We hypothesis that sirolimus coated balloon is superior to conventional plain balloon angioplasty with decreased re-stenosis of target lesion, improved access circuit and target lesion patency, and decreased number of interventions needed to maintain patency.

DETAILED DESCRIPTION:
Dialysis vascular accesses such as Arteriovenous Fistula (AVF) and Arteriovenous Grafts (AVG) are surgically created vasculatures used for hemodialysis in patients with End Stage Renal Disease (ESRD). A functioning dialysis vascular access is critical to the delivery of life-saving hemodialysis (HD) treatment to these patients. Unfortunately, neointimal hyperplasia frequently occurs within the dialysis vascular access, resulting in stenosis, poor flow and thrombosis with loss of function. The durability of both AVF and AVG are poor, with an almost 50% failure rate after a median lifetime of 3 to 7 years for AVF and 12 to 18 months for AVG. Vascular access failure is the most common reason for hospitalization among HD patients. The global healthcare costs for treating vascular access-related complications amount to USD 18 billion, and in USD 1 billion in the US alone. These figures are set to increase, due to the increase in prevalence of access interventions and hemodialysis patients globally. Singapore has one of the highest ESRD rates in the world and investigators are facing an increasing number of patients with ESRD and majority of the patients opting for hemodialysis as their treatment modality. As such, vascular access related complication is set to be a major contribution of healthcare cost in our nation.

Thrombosis of dialysis access is a catastrophic event in patients with ESRD as it results in a loss of access to hemodialysis. Thrombosis is often as a result of underlying stenosis in the dialysis circuit. To restore the function of the dialysis access, the thrombus is lysed with the use of lytic agents; followed by treatment of the underlying stenosis. The current gold standard therapy for treatment of stenosis in dialysis access is plain balloon angioplasty (BA). Despite its widespread availability and minimally invasive nature, the mid- and long-term patency with BA in patients with ESRD is poor. The reported average primary patency after BA is around 40-50% at 1 year. Multiple repeated angioplasty are required to maintain the patency of the vascular access. Hence, there is an urgent clinical need to improve the patency of dialysis vascular access.

Recently, the use of stents, in particular stent graft, has been shown to be superior to angioplasty for stenosis occurring at the site of venous anastomoses of an AVG. The incidence of patency of the treatment area was significantly greater in the stent-graft group than in the balloon-angioplasty group (51% vs. 23%, P<0.001), as was the incidence of patency of the access circuit (38% vs. 20%, P=0.008) at 6 months. For cephalic arch stenosis in AVF, the use of stent graft has also been shown to be superior to bare metal stent. The 6 month primary patency for stent graft and bare stent was 81.8 and 39.1%, respectively. One-year primary patency for stent graft and bare stent was 31.8 and 0.00%, respectively (P = 0.002). However, the use of stent graft for the management of dialysis vascular access is not without any concern. In particular, re-stenosis can occur within the stented segment (post stent 12-month primary patency is 46%), resulting in the need for repeat angioplasty. Future stent deployment in the re-stenotic segment may also not be feasible due to the presence of the stent. Moreover, the presence of a stent can impede future surgical revision or new access creation within the same vessel.

Paclitaxel-coated balloon angioplasty (PCBA) has also been shown recently to be superior to plain BA in the treatment of stenosis in dialysis vascular access. This is because the very intervention used to treat the underlying stenosis by plain BA can induce vascular injury and accelerate intimal hyperplasia, resulting in rapid restenosis and need for repeated procedures to maintain vessel patency. By releasing Paclitaxel, which is an anti-proliferative drug, locally into the vessel wall during balloon contact, it will blunt the acceleration of intimal hyperplasia response, resulting in improved primary patency after angioplasty. Additionally, unlike stents, PCBA does not leave a permanent structure that may impede future surgical revision. In a small 40 patient pilot study, the primary unassisted patency in the PCBA group was significantly better than the plain BA group at 6 (70 % versus 25 %) and 12 months (35 % versus 5 %, p <0.001) respectively.

Sirolimus coated balloon (SCB) is the new generation of drug eluting balloons that are available in the market. Compared to Paclitaxel, sirolimus is cytostatic in its mode of action with a high margin of safety. It has a high transfer rate to the vessel wall and effectively inhibit neointimal hyperplasia in the porcine coronary model. In the coronary artery interventions, preliminary clinical studies using SCB have also shown excellent procedural and 6 month patency.

The effectiveness of SCB in patients with dialysis access dysfunction has not been previously investigated. As thrombosis frequently occur as a result of underlying stenosis from neointimal hyperplasia, investigators postulate that the application of SCB after successful thrombolysis will inhibit the onset of neointimal hyperplasia and result in better vascular access patency. Specifically for AVG, where thrombosis episodes are frequent and the 3 month patency rate after successful thrombolysis is only 40%, investigators hypothesize that the application of SCB after successful thrombolysis in AVG may be the key to improving the mid and long term patency of the AVG after successful thrombolysis.

Investigators intended to perform this single centre study with a planned total of 20 patients enrolled from Singapore General Hospital. The patient pool will be from adult renal failure patients with successfully thrombolysis of thrombosed AVG admitted to SGH between June 2018 and December 2018. Adult patients of both genders and all races may be included in this study. Children and pregnant women will not be included in this study as they are considered a vulnerable population and are also not representative of the population at risk.

Patients who are admitted to the hospital for thrombosed AVG will be screened and offered enrollment if they meet the inclusion criteria. Patients will be consented and pre-procedure blood tests (full blood count, renal panel and PT/PTT) performed as per standard hospital criteria. Patients who have successful thrombolysis will be recruited into the study and receive the sirolimus coated balloon in the same setting. Patients who have unsuccessful thrombolysis will be considered as screen failures and will not be recruited into the trial.

Thrombolysis of the AVG will be performed as per standard hospital protocol in the Interventional Nephrology suite (INS). Briefly, an antegrade and retrograde vascular sheath will be placed in the thrombosed AVG under ultrasound guidance. Thrombolytic agents will be delivered into the thrombosed AVG via the vascular sheaths or infusion catheters. The culprit venous stenosis will be treated using plain BA and thrombus within the AVG macerated using the same angioplasty balloon. The arterial plug will be dislodged by using a 5.5Fr Fogarty balloon. Following successful thrombolysis of the AVG, the number and location of lesions within the dialysis circuit will be documented. After adequate angioplasty of the culprit lesion (defined as <30% residual stenosis after treatment at rated burst pressure of the angioplasty balloon), SCB will be applied at the culprit lesion after appropriate sizing using the diameter of the graft or the outflow vein as reference. To ensure adequate contact, the SCB should be of the same or oversized by 1mm the diameter of the reference vessel. An inflation device with a pressure gauge will be used to inflate up to manufacturers' stated burst pressure. The duration of balloon inflation will be 2 minutes at the rated burst pressure. Post angioplasty with SCB, a completion graftogram will be done to document the results. The size of the balloon used, inflation pressure, the transit time of balloon, number of inflation, procedure complications (if any), and residual stenosis will be recorded.

Post procedure, all patients will received daily dose aspirin (100mg) and clopidogrel (75mg) orally for 1 month, followed by treatment with aspirin alone for 6 months. For patients who are already on Aspirin prior to the procedure, they will continue on aspirin after the trial. For patients who are already on clopidogrel before the trial, they will continue on clopidogrel after 1 month of combination therapy with aspirin.

As patients with ESRD are at increased risk of bleeding, proton pump inhibitors will be prescribed during the period that they are receiving dual anti-platelet therapy. Patients will also be informed of the risk of bleeding and to seek immediate medical attention should they develop any bleeding episodes. The patients will be followed up via monthly phone call from the principle investigator while they are on dual anti-platelet therapy.

Investigators define patency based on SIR reporting standards (Gray et al., 2003):

Post-intervention target lesion patency:

Interval after intervention until the next re-intervention at or adjacent to the original treatment site or until the access is abandoned. Percutaneous or surgical treatments of a new arterial or venous outflow stenosis/occlusion (including access thrombosis) that do not involve or exclude the original lesion from the access circuit are compatible with lesion patency. Creation of a new access that incorporates the target lesion into the new access circuit is also compatible with target lesion patency.

Post-intervention access circuit primary patency:

Interval following intervention until the next access thrombosis or repeated intervention. It ends with the treatment of a lesion anywhere within the access circuit, from the arterial inflow to the superior vena cava-right atrial junction.

Post-intervention access circuit assisted primary patency:

Interval after intervention until access thrombosis or a surgical intervention that excludes the treated lesion from the access circuit. Percutaneous treatments of either restenosis/occlusion of the previously treated lesion or a new arterial or venous outflow stenosis/occlusion (excluding access thrombosis) are compatible with assisted primary patency.

Post-intervention access circuit secondary patency:

Interval after intervention until the access is surgically declotted, revised or abandoned. Thrombolysis and percutaneous thrombectomy are compatible with secondary patency.

With regards to the potential complication, it will be categorised according to SIR definitions of minor or major complications (Aruny et al., 2003):

A major complication is defined as one that:

1. require therapy, minor hospitalisation (< 48 hours),
2. require major therapy, unplanned increase in level of care, prolonged hospitalisation (>48 hours),
3. leads to permanent adverse sequelae, or
4. death

A minor complication is one that:

1. requires no therapy with no consequence,
2. requires nominal therapy with no consequence; includes overnight admission for observation only.

All participants will be followed-up after intervention to assess the patency clinically and radiologically as well as complications and whether able to achieve prescribed haemodialysis.

All participants will be received call from principal investigator or site-investigator or study members monthly to assess the compliance to antiplatelet therapy as well as assess whether any adverse effects associated with antiplatelet therapy.

The participant is seen for assessment of primary outcome. The window period for this scheduled post-intervention visit is 3 month post-intervention ± 1 weeks.

The participant returns for a 6-month follow-up to assess the patency rate of AVG as well as any intervention needed to maintain patency.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-85 years
2. Thrombosed AVG in the arm
3. Successful thrombolysis of the thrombosed AVG, defined as the re-established of flow on Digital Subtraction Angiography (DSA) and restoration of thrill in the AVG on clinical examination

Exclusion Criteria:

1. Patient unable to provide informed consent
2. Previous bare metal stent or stent-graft placement within the dialysis access
3. Presence of central vein stenosis
4. Sepsis or active infection
5. Recent intracranial bleed or gastrointestinal bleed within the past 12 months
6. Allergy to iodinated contrast media, anti-platelet drugs, heparin or paclitaxel
7. Pregnancy
8. Life expectancy < 12 months based on physician's estimate (active malignancy)

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
The patency rate of AVG at 3 months post sirolimus balloon angioplasty by performing surveillance ultrasound of AVG, assessing the thrill of AVG and assessing any dysfunctional vascular assess- related hospital admission. | 3 months

SECONDARY OUTCOMES:
The patency rate of AVG at 6 months post sirolimus balloon angioplasty by performing surveillance ultrasound of AVG, assessing the thrill of AVG and assessing any dysfunctional vascular assess- related hospital admission. | 6 months
The number of intervention(s) needed to maintain patency of AVG. | 6 months
The cost effective of using sirolimus coated balloon in the management of thrombosed AVG by reviewing hospital bills related to dysfunctional dialysis access. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Chieh Suai Tan, Doctor, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital Renal Department, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roy-Chaudhury P, Sukhatme VP, Cheung AK. Hemodialysis vascular access dysfunction: a cellular and molecular viewpoint. J Am Soc Nephrol. 2006 Apr;17(4):1112-27. doi: 10.1681/ASN.2005050615. PMID 16565259
- [Background] Lee T, Roy-Chaudhury P. Advances and new frontiers in the pathophysiology of venous neointimal hyperplasia and dialysis access stenosis. Adv Chronic Kidney Dis. 2009 Sep;16(5):329-38. doi: 10.1053/j.ackd.2009.06.009. PMID 19695501
- [Result] Pantelias K, Grapsa E. Vascular access today. World J Nephrol. 2012 Jun 6;1(3):69-78. doi: 10.5527/wjn.v1.i3.69. PMID 24175244
- [Result] Collins AJ, Foley RN, Gilbertson DT, Chen SC. United States Renal Data System public health surveillance of chronic kidney disease and end-stage renal disease. Kidney Int Suppl (2011). 2015 Jun;5(1):2-7. doi: 10.1038/kisup.2015.2. PMID 26097778
- [Result] Rajan DK, Bunston S, Misra S, Pinto R, Lok CE. Dysfunctional autogenous hemodialysis fistulas: outcomes after angioplasty--are there clinical predictors of patency? Radiology. 2004 Aug;232(2):508-15. doi: 10.1148/radiol.2322030714. PMID 15286321
- [Result] Manninen HI, Kaukanen ET, Ikaheimo R, Karhapaa P, Lahtinen T, Matsi P, Lampainen E. Brachial arterial access: endovascular treatment of failing Brescia-Cimino hemodialysis fistulas--initial success and long-term results. Radiology. 2001 Mar;218(3):711-8. doi: 10.1148/radiology.218.3.r01mr38711. PMID 11230644
- [Result] Heye S, Maleux G, Vaninbroukx J, Claes K, Kuypers D, Oyen R. Factors influencing technical success and outcome of percutaneous balloon angioplasty in de novo native hemodialysis arteriovenous fistulas. Eur J Radiol. 2012 Sep;81(9):2298-303. doi: 10.1016/j.ejrad.2011.09.004. Epub 2011 Sep 28. PMID 21955605
- [Result] Haskal ZJ, Trerotola S, Dolmatch B, Schuman E, Altman S, Mietling S, Berman S, McLennan G, Trimmer C, Ross J, Vesely T. Stent graft versus balloon angioplasty for failing dialysis-access grafts. N Engl J Med. 2010 Feb 11;362(6):494-503. doi: 10.1056/NEJMoa0902045. PMID 20147715
- [Result] Shemesh D, Goldin I, Zaghal I, Berlowitz D, Raveh D, Olsha O. Angioplasty with stent graft versus bare stent for recurrent cephalic arch stenosis in autogenous arteriovenous access for hemodialysis: a prospective randomized clinical trial. J Vasc Surg. 2008 Dec;48(6):1524-31, 1531.e1-2. doi: 10.1016/j.jvs.2008.07.071. Epub 2008 Oct 1. PMID 18829240
- [Result] Katsanos K, Karnabatidis D, Kitrou P, Spiliopoulos S, Christeas N, Siablis D. Paclitaxel-coated balloon angioplasty vs. plain balloon dilation for the treatment of failing dialysis access: 6-month interim results from a prospective randomized controlled trial. J Endovasc Ther. 2012 Apr;19(2):263-72. doi: 10.1583/11-3690.1. PMID 22545894
- [Result] Andreini D, Trabattoni D. Is the Sirolimus encapsulated balloon a reliable tool for treating the in-stent restenosis?-insights from the SABRE trial. J Thorac Dis. 2018 Feb;10(2):634-637. doi: 10.21037/jtd.2018.01.05. No abstract available. PMID 29607127
- [Result] Verheye S, Vrolix M, Kumsars I, Erglis A, Sondore D, Agostoni P, Cornelis K, Janssens L, Maeng M, Slagboom T, Amoroso G, Jensen LO, Granada JF, Stella P. The SABRE Trial (Sirolimus Angioplasty Balloon for Coronary In-Stent Restenosis): Angiographic Results and 1-Year Clinical Outcomes. JACC Cardiovasc Interv. 2017 Oct 23;10(20):2029-2037. doi: 10.1016/j.jcin.2017.06.021. Epub 2017 Sep 27. PMID 28964764
- [Derived] Tan RY, Tan CW, Pang SC, Foo MWY, Tang TY, Gogna A, Chong TT, Tan CS. Study protocol of a pilot study on sirolimus-coated balloon angioplasty in salvaging clotted arteriovenous graft. CVIR Endovasc. 2020 Jul 5;3(1):34. doi: 10.1186/s42155-020-00123-4. PMID 32627114